CLINICAL TRIAL: NCT03420378
Title: Central Sensitization in Vitamin D Deficiency and Effect of Vitamin D Replacement on Cutaneous Silent Period
Brief Title: Central Sensitization in Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12.2017.123
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Vitamin D Deficiency; Central Sensitisation
Keywords: Central Sensitisation; Cutaneous Silent Period; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): Patients with vitamin D deficiency will receive vitamin D replacement therapy. Before and after therapy, cutaneous silent period will be measured from each upper extremity and latencies will be recorded. Their LANSS scores and Notthingham Health Profile will be recorded before and after treatment.
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — Vitamin D replacement

SUMMARY:
The purpose of this study is to investigate the presence of central sensitization in vitamin D deficiency and its effect on cutaneous silent period, pain, and quality of life. The secondary purpose of the study is to investigate whether a change in cutaneous silent period parameters, pain severity and neuropathic sensitization and quality of life after vitamin D replacement.

DETAILED DESCRIPTION:
Vitamin D deficiency is a pandemia. Main causes of this is insufficient exposure to sunlight. Vitamin D deficiency is related to conditions like various cancers, autoimmune diseases, hypertension and growth retardation in children (1).

International Association for the study of pain has defined pain as "An unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage." (2). Pain lasting longer than 3 months has been deemed as chronic pain (3). Vitamin D deficiency influences various types of pain, including chronic pain (4,5,6,7).

Vitamin D influences the musculoskeletal system via the calcium-phosphorus metabolism and the receptors found in skeletal muscle cells (8). Vitamin D deficiency has been shown to decrease muscle strength, the this decrease in proximal muscles affect postural stability and can increase falls. Vitamin D deficiency also causes problems in bone mineralization, causing isolated or widespread pain in muscles, bones and joints. These patients end up getting wrong diagnoses such as fibromyalgia, osteoarthritis, inflammatory arthritis, and chronic fatigue syndrome (1,7). Vitamin D deficiency causes hyperinnervation and hypersensitivity on nerves and cause pain to be felt more intensely (5).

In a normal skeletal muscle, during an isometric contraction, a number of motor unit will be activated. These motor units produce a stable electromyography pattern and keep their own frequencies during contraction. If the nerve, tendon or a cutaneous nerve nearby is stimulated, electromyographic activity is disrupted and a bioelectric silence occurs. This is called cutaneous silent period (CSP). It is an inhibitory spinal reflex and its afferents consist of A-delta nerve fibers.

In various studies, CSP has been shown to be clinically beneficial in conditions like peripheral neuropathy, syringomyelia, Parkinson's disease, restless leg syndrome and fibromyalgia.

von Känel R et al. has investigated the effect of vitamin D deficiency on widespread pain index (WPI) and symptom severity score (SSS) and found out that it increases central sensitivity (8). In thei study, thy did not utilize any electrophysiologic objective measurements. Akyüz et al. have investigated the effect of vitamin D deficiency on chronic pain and nerve conduction studies; they have shown that vitamin D is correlated with various nerve conduction parameters while these parameters do not change after replacement (9,10).

Patients with vitamin D deficiency and healthy controls with normal vitamin D levels will be compared in terms of cutaneous silent period parameters, pain severity and neuropathic sensitization and quality of life. Cutaneous silent period parameters (duration and latency ), The Leeds Assessment of Neuropathic Symptoms & Signs and Nottingham Health Profile will be used for the assessments. Patients with vitamin D deficiency will receive vitamin D supplementation therapy. Before and after therapy, cutaneous silent period parameters, LANSS scores and Nottingham Health Profile will measured before and 8 weeks after starting vitamin D supplementation therapy.

ELIGIBILITY:
Inclusion Criteria

* Presence of widespread pain
* Presence of vitamin D deficit

Exclusion Criteria:

* Any contraindication of performing silent cutaneous period
* Any contraindication for vitamin d use
* Presence of conditions that affect cutaneous silent period like the presence of carpal tunnel syndrome and polyneuropathies
* Defective peripheric autonomic nervous system findings
* Not being able to write and read
* Not being able to communicate

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
cutaneous silent period latency (ms) | 8 weeks
  the brief interruption in voluntary contraction that follows strong electrical stimulation (painful) of a cutaneous nerve
cutaneous silent period duration (ms) | 8 weeks
  the brief interruption in voluntary contraction that follows strong electrical stimulation (painful) of a cutaneous nerve

SECONDARY OUTCOMES:
Visual analog scale (VAS) of pain | 8 weeks
  line from 0: no pain to 10:worst pain
Leeds assessment of neuropathic symptoms and signs (LANSS) | 8 weeks
  Reduction of pain related to central sensitization. LANSS scale ⩾ 12 refers to "Neu- neuropathic sensitization"
The Nottingham Health Profile (NHP) | 8 weeks
  The Nottingham Health Profile is intended for primary health care, to provide a brief indication of a patient's perceived emotional, social and physical health problems. The number of questions answered "yes" in each subgroup is divided by the total number of questions in the same subgroup and the result is multiplied by 100. Each subgroup has a value of between 0 and 100, with 100 points being considered the best general QoL for the calculated subgroup and 0 points being considered as the worst QoL for the same subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Kenis Coskun, MD, Principal Investigator — Marmara Universtiy
Locations (1):
- Ozge Kenis Coskun, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF. Vitamin D: importance in the prevention of cancers, type 1 diabetes, heart disease, and osteoporosis. Am J Clin Nutr. 2004 Mar;79(3):362-71. doi: 10.1093/ajcn/79.3.362. PMID 14985208
- [Background] Hamilton B. Vitamin D and human skeletal muscle. Scand J Med Sci Sports. 2010 Apr;20(2):182-90. doi: 10.1111/j.1600-0838.2009.01016.x. Epub 2009 Oct 5. PMID 19807897
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Lotfi A, Abdel-Nasser AM, Hamdy A, Omran AA, El-Rehany MA. Hypovitaminosis D in female patients with chronic low back pain. Clin Rheumatol. 2007 Nov;26(11):1895-901. doi: 10.1007/s10067-007-0603-4. Epub 2007 Mar 22. PMID 17377737
- [Background] Wicherts IS, van Schoor NM, Boeke AJ, Visser M, Deeg DJ, Smit J, Knol DL, Lips P. Vitamin D status predicts physical performance and its decline in older persons. J Clin Endocrinol Metab. 2007 Jun;92(6):2058-65. doi: 10.1210/jc.2006-1525. Epub 2007 Mar 6. PMID 17341569
- [Background] Mascarenhas R, Mobarhan S. Hypovitaminosis D-induced pain. Nutr Rev. 2004 Sep;62(9):354-9. doi: 10.1111/j.1753-4887.2004.tb00061.x. PMID 15497769
- [Background] Gloth FM 3rd, Lindsay JM, Zelesnick LB, Greenough WB 3rd. Can vitamin D deficiency produce an unusual pain syndrome? Arch Intern Med. 1991 Aug;151(8):1662-4. PMID 1872673
- [Background] Haroon M, FitzGerald O. Vitamin D deficiency: subclinical and clinical consequences on musculoskeletal health. Curr Rheumatol Rep. 2012 Jun;14(3):286-93. doi: 10.1007/s11926-012-0244-8. PMID 22328176
- [Background] Tague SE, Clarke GL, Winter MK, McCarson KE, Wright DE, Smith PG. Vitamin D deficiency promotes skeletal muscle hypersensitivity and sensory hyperinnervation. J Neurosci. 2011 Sep 28;31(39):13728-38. doi: 10.1523/JNEUROSCI.3637-11.2011. PMID 21957236
- [Background] von Kanel R, Muller-Hartmannsgruber V, Kokinogenis G, Egloff N. Vitamin D and central hypersensitivity in patients with chronic pain. Pain Med. 2014 Sep;15(9):1609-18. doi: 10.1111/pme.12454. Epub 2014 Apr 14. PMID 24730754
- [Background] Kuru P, Akyuz G, Yagci I, Giray E. Hypovitaminosis D in widespread pain: its effect on pain perception, quality of life and nerve conduction studies. Rheumatol Int. 2015 Feb;35(2):315-22. doi: 10.1007/s00296-014-3099-7. Epub 2014 Aug 2. PMID 25085713
- [Background] Akyuz G, Sanal-Toprak C, Yagci I, Giray E, Kuru-Bektasoglu P. The effect of vitamin D supplementation on pain, quality of life, and nerve conduction studies in women with chronic widespread pain. Int J Rehabil Res. 2017 Mar;40(1):76-83. doi: 10.1097/MRR.0000000000000211. PMID 28030514